CLINICAL TRIAL: NCT05789719
Title: An Exploratory Clinical Study to Investigate the Effect of autoSTEM-OA and alloSTEM-OA in Participants With Knee Osteoarthritis.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: StemMedical A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ST-001
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- autoSTEM-OA 400 (Experimental): 400x10^6 autologous MSC(AT)s in autologous fat
  Interventions: Biological: STEM-OA
- alloSTEM-OA 400 (Experimental): 400x10^6 allogeneic MSC(AT)s in autologous fat
  Interventions: Biological: STEM-OA
- autoSTEM-OA 800 (Experimental): 800x10^6 autologous MSC(AT)s in autologous fat
  Interventions: Biological: STEM-OA
- alloSTEM-OA 800 (Experimental): 800x10^6 allogeneic MSC(AT)s in autologous fat
  Interventions: Biological: STEM-OA
- autoSTEM-OA 1600 (Experimental): 1600x10^6 autologous MSC(AT)s in autologous fat
  Interventions: Biological: STEM-OA
- alloSTEM-OA 1600 (Experimental): 1600x10^6 allogeneic MSC(AT)s in autologous fat
  Interventions: Biological: STEM-OA

INTERVENTIONS:
Biological: STEM-OA — Combination of autologous or allogeneic MSC(AT)s and fat

SUMMARY:
A phase 1 exploratory clinical study to investigate safety, tolerance and efficacy of a single intra-articular injection of autoSTEM-OA or alloSTEM-OA in participants with mild to moderate knee osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
2. Male or female, aged 18 - 60 years (both inclusive) at the time of informed consent.
3. Joint pain ≥ 30mm on 100mm VAS at screening
4. Grade 2-3 Kellgren Lawrence OA on radiograph with no full-thickness lesion >1 cm in any dimension by x-ray
5. Failure of minimum 2 nonoperative therapies (oral pain medications, physical therapy, corticosteroid injection, or viscosupplementation injection)
6. Body mass index (BMI) within the range 18 - 35 kg/m2 (both inclusive)
7. Minimum 200 ml of fat (lipoaspirate) available for liposuction at the abdomen and/or thighs as judged by the investigator.
8. Agree to donate cells to alloSTEM-OA participants.
9. Fulfils eligibility criteria for allogeneic cell- and tissue donors.
10. Speaks and reads Danish or English

Exclusion Criteria:

1. Active tobacco use, or use of other nicotine substitutes
2. Active cancer or still in follow-up (5 years)
3. Rheumatologic disease
4. Avascular disease
5. Severe bone deformity
6. Previous infection of the knee joint
7. Pes anserine bursitis
8. pain attributed to diffuse edema
9. pain attributed to displaced meniscal tear or osteochondritis
10. Neurogenic or vascular claudication
11. Bleeding disorders
12. Chemotherapy
13. Radiation therapy to the leg or adipose harvested site
14. Knee injections within 3 months of treatment
15. Unable to discontinue the following drugs 7 days before injections (prescription pain medication, anticoagulation medicine (including ibuprofen), thrombolytics, antiplatelet medication)
16. Use of oral glucocorticoids.
17. Female who is pregnant, breast-feeding or intends to become pregnant within 1-year after the treatment, or is of child-bearing potential and not using highly effective contraceptive method.
18. Known chronic disease associated with metabolism malfunction or poor healing.
19. Allergy towards necessary anaesthesia
20. Varus/valgus malalignment >5°
21. Isolated patellofemoral arthrosis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
STEM-OA safety | 13 weeks
  Number of treatment emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Knee pain | 13 weks
  Change in KOOS 'pain' score
Number of treatment responders | 13 weks
  Number of treatment responders according to the OMERACT-OARSI criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Sanos Clinic Syddanmark, Vejle, Denmark

IPD SHARING:
Plan to Share IPD: Undecided